CLINICAL TRIAL: NCT06550167
Title: Neuroprotective Effect of Omega (Nano PSO), Changes in Neurotrophic BDNF and VEGF, and Their Association With Cognitive Status in Patients Who Used to Consume Psychoactive Substances
Brief Title: Neuroprotective Effect of (Nano PSO), in Patients Who Used to Consume Psychoactive Substances
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Distribuidora Biolife SA de CV (Industry)
Responsible Party: Principal Investigator, Irene Guadalupe Aguilar García, Principal Investigator,, Distribuidora Biolife SA de CV
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-122
Record Dates: First submitted 2024-06-13; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Addiction;Drug(S);LSD; Neuroprotective
Keywords: Addiction, Drug; Neuroprotective; pomegranate seed oil
MeSH Terms: conditions — Substance-Related Disorders | interventions — Nano-PSO; Nanotechnology

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The randomized drawing was carried out through the Randomization.com program, which is an online platform that provides randomization services for clinical studies.
  In addition, the treatments received were previously labeled and randomized by the sponsor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nano-PSO (Experimental): Nano-PSO or Pomegranate seed oil with nanotechnology, capsules with a net content of 640mg with a dosage indicated by sponsor of 2 capsules in fast
  Interventions: Dietary Supplement: Nano-PSO, Pomegranate seed oil (omega-5)
- PLACEBO (Placebo Comparator): Placebo physically identical to Nano-PSO capsules Soft gelatin capsules 640 mg edible oil for PLACEBO being the following information: oil edible, oval shape, 640 mg
  Interventions: Other: PLACEBO

INTERVENTIONS:
Dietary Supplement: Nano-PSO, Pomegranate seed oil (omega-5) — During the intervention, Nano-PSO dietary supplement will be administered to the participants in the assigned group.
  Participants will be followed before and after treatment to assess the effects of Nano-PSO on cognitive status, serum concentrations of trophic factors, and other relevant parameters . This randomized, double-blind, controlled clinical trial design allows for a rigorous evaluation of the potential benefits of Nano-PSO in patients with substance use disorders. The study aims to provide valuable insights into the neuroprotective and cognitive-enhancing properties of Nano-PSO in this population.
  Other Names: Oil of pomegranate seed with nanotechnology
  Arms: Nano-PSO
Other: PLACEBO — In this arm of the study the participants will receive a placebo as a control treatment . The placebo is essential in clinical trials to compare the effects of the active intervention (Nano-PSO) with those of an inert substance.
  Arms: PLACEBO

SUMMARY:
Addiction problems to psychoactive substances are becoming more frequent, which implies a serious health problem, with social, family and work repercussions. Participants with chronic consumption present important degeneration processes mediated by Neuroinflammation, oxidative stress and excitotoxicity. At the moment there is no effective treatment that can reduce the damage. The effectiveness of Omega 5 has been demonstrated in different disorders of the nervous system; However, very little has been elucidated about the mechanisms of regulation and activation in consumer patients. Omega 5 Nano-PSO has an important role in mechanisms of cell survival in different pathological events.

In this project aims to explain the possible mechanisms underlying the morphological changes and pathologies associated with oxidative stress and inflammation, since it could be a useful strategy to counteract the effects of substances of abuse on brain cells.

Omega 5 (Nano PSO) will modify the levels of neurotrophic factors through the decrease in inflammation and reactive oxygen species in patient-consumers of substances, reducing neuronal death and therefore cognitive deterioration. Methodological design Type of study: Clinical trial, randomized controlled, double blind. Research Headquarters: This work will be carried out at the University Center for Health Science with the participation of the "My family is waiting for me" rehabilitation centers. Study Period: 2 years

DETAILED DESCRIPTION:
Omega 5 (Nano PSO) has been shown to be a powerful antioxidant with neuroprotective and anti-inflammatory effects in various neurological and neurodegenerative diseases. In patients who consume psychoactive substances, who present high levels of neuroinflammation and oxidative stress, Omega 5 could help to reduce damage on neuronal and glial cells, promoting cell survival and preserving a homeostatic microenvironment in the brain.

It has been suggested that Omega 5 could modify the levels of neurotrophic factors such as BDNF and VEGF, which might contribute to the protection of brain cells and the improvement of cognitive status in substance abuse patients. In addition, it has been mentioned that Omega 5 acts through the reduction of inflammation and reactive oxygen species, which could reduce neuronal death and prevent cognitive deterioration in these patients.

In summary, Omega 5 (Nano PSO) seems to play an important role in protecting the brain cells of patients who consume psychoactive substances by acting as an antioxidant and anti-inflammatory, modulating neurotrophic factors and promoting cell survival in a brain environment affected by substance consumption.

It has been investigated that Omega 5 (Nano PSO) exerts its beneficial effects through various regulation and activation mechanisms in patients who consume psychoactive substances:

1. Modulation of neurotrophic factors: It has been suggested that Omega 5 can modify the levels of neurotrophic factors such as brain-derived neurotrophic factor (BDNF) and vascular endothelial growth factor (VEGF) in patients who consume psychoactive substances. These factors play a crucial role in the neuroprotection, and its modulation by Omega 5 could contribute to the improvement of cognitive status and cell survival in these patients.
2. Antioxidant and anti-inflammatory action: Omega 5 has been shown to have antioxidant and anti-inflammatory effects in several pathologies of the nervous system. In patients who consume psychoactive substances, who have high levels of neuroinflammation and oxidative stress, Omega 5 can help reduce damage to neuronal and glial cells, promoting cell survival and preserving a homeostatic brain environment.
3. Protection against oxidative stress: It has been suggested that Omega 5 may be useful to reduce the damage caused by oxidative stress at the brain level in substance abuse patients. By acting as an antioxidant, Omega 5 could counteract the negative effects of oxidative stress on brain cells and contribute to neuronal protection.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are multiple users of methamphetamines, cocaine, and cannabis with or without alcohol and tobacco, and have a history of at least 3 years of consumption.
* Patients who accept informed consent to participate in the protocol.
* Male gender.
* Age between 18-50 years in the withdrawal phase currently in residential treatment

Exclusion Criteria:

* Individuals under 18 years of age.
* Patients who do not sign the informed consent.
* Discharge of patients prior to the stipulated 6 months, requested by family members.
* Patients with developed or known allergies.
* Patients who are consuming NSAIDs, MAOIs (monoamine oxidase Inhibitor), active chronic inflammatory diseases, or any type of cancer

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Serum Brain-derived neurotrophic factor (BDNF) and Vascular endothelial growth factor VEGF Concentrations after treatment | A BASELINE EVALUATION AND AN EVALUATION AFTER SIX MONTHS OF INTERVENTION
  ELISA kittesting will be performed on blood samples to measure BDNF and VEGF concentrations before and after Nano PSO treatment.

SECONDARY OUTCOMES:
Changes in the Montreal Cognitive Assessment (MoCA) after treatment. | A BASELINE EVALUATION AND AN EVALUATION AFTER SIX MONTHS OF INTERVENTION
  A neuropsychological battery will be designed to evaluate different cognitive aspects and the results of (Montreal Cognitive Assessment (MoCA) obtained will be interpreted.

CONTACTS AND LOCATIONS:
Overall Officials: Irene G Aguilar, PH, Principal Investigator — University of Guadalajara
Locations (1):
- Irene Guadalupe Aguilar García PhD., Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdel-Zaher AO, Mostafa MG, Farghly HM, Hamdy MM, Omran GA, Al-Shaibani NK. Inhibition of brain oxidative stress and inducible nitric oxide synthase expression by thymoquinone attenuates the development of morphine tolerance and dependence in mice. Eur J Pharmacol. 2013 Feb 28;702(1-3):62-70. doi: 10.1016/j.ejphar.2013.01.036. Epub 2013 Jan 30. PMID 23376567
- [Result] Abdel-Zaher AO, Mostafa MG, Farghaly HS, Hamdy MM, Abdel-Hady RH. Role of oxidative stress and inducible nitric oxide synthase in morphine-induced tolerance and dependence in mice. Effect of alpha-lipoic acid. Behav Brain Res. 2013 Jun 15;247:17-26. doi: 10.1016/j.bbr.2013.02.034. Epub 2013 Mar 5. PMID 23470902
- [Result] Adu-Frimpong M, Firempong CK, Omari-Siaw E, Wang Q, Mukhtar YM, Deng W, Yu Q, Xu X, Yu J. Preparation, optimization, and pharmacokinetic study of nanoliposomes loaded with triacylglycerol-bound punicic acid for increased antihepatotoxic activity. Drug Dev Res. 2019 Mar;80(2):230-245. doi: 10.1002/ddr.21485. Epub 2018 Nov 10. PMID 30414214
- [Result] Andreska T, Aufmkolk S, Sauer M, Blum R. High abundance of BDNF within glutamatergic presynapses of cultured hippocampal neurons. Front Cell Neurosci. 2014 Apr 11;8:107. doi: 10.3389/fncel.2014.00107. eCollection 2014. PMID 24782711
- [Result] Aruna P, Venkataramanamma D, Singh AK, Singh RP. Health Benefits of Punicic Acid: A Review. Compr Rev Food Sci Food Saf. 2016 Jan;15(1):16-27. doi: 10.1111/1541-4337.12171. Epub 2015 Oct 21. PMID 33371578
- [Result] Berrios-Carcamo P, Quezada M, Quintanilla ME, Morales P, Ezquer M, Herrera-Marschitz M, Israel Y, Ezquer F. Oxidative Stress and Neuroinflammation as a Pivot in Drug Abuse. A Focus on the Therapeutic Potential of Antioxidant and Anti-Inflammatory Agents and Biomolecules. Antioxidants (Basel). 2020 Sep 4;9(9):830. doi: 10.3390/antiox9090830. PMID 32899889
- [Result] Castillo-Navarrete JL, Guzman-Castillo A, Bustos C, Rojas R. Peripheral brain-derived neurotrophic factor (BDNF) and salivary cortisol levels in college students with different levels of academic stress. Study protocol. PLoS One. 2023 Feb 22;18(2):e0282007. doi: 10.1371/journal.pone.0282007. eCollection 2023. PMID 36812175
- [Result] Cai Y, Yang L, Hu G, Chen X, Niu F, Yuan L, Liu H, Xiong H, Arikkath J, Buch S. Regulation of morphine-induced synaptic alterations: Role of oxidative stress, ER stress, and autophagy. J Cell Biol. 2016 Oct 24;215(2):245-258. doi: 10.1083/jcb.201605065. Epub 2016 Oct 17. PMID 27810915
- [Result] Famitafreshi H, Karimian M. Socialization Alleviates Burden of Oxidative-Stress in Hippocampus and Prefrontal Cortex in Morphine Addiction Period in Male Rats. Curr Mol Pharmacol. 2018;11(3):254-259. doi: 10.2174/1874467210666170919161045. PMID 28933310
- [Result] George O, Koob GF. Individual differences in prefrontal cortex function and the transition from drug use to drug dependence. Neurosci Biobehav Rev. 2010 Nov;35(2):232-47. doi: 10.1016/j.neubiorev.2010.05.002. Epub 2010 May 20. PMID 20493211
- [Result] Guerra-Vazquez CM, Martinez-Avila M, Guajardo-Flores D, Antunes-Ricardo M. Punicic Acid and Its Role in the Prevention of Neurological Disorders: A Review. Foods. 2022 Jan 18;11(3):252. doi: 10.3390/foods11030252. PMID 35159404
- [Result] Guillin O, Diaz J, Carroll P, Griffon N, Schwartz JC, Sokoloff P. BDNF controls dopamine D3 receptor expression and triggers behavioural sensitization. Nature. 2001 May 3;411(6833):86-9. doi: 10.1038/35075076. PMID 11333982
- [Result] Grimm JW, Lu L, Hayashi T, Hope BT, Su TP, Shaham Y. Time-dependent increases in brain-derived neurotrophic factor protein levels within the mesolimbic dopamine system after withdrawal from cocaine: implications for incubation of cocaine craving. J Neurosci. 2003 Feb 1;23(3):742-7. doi: 10.1523/JNEUROSCI.23-03-00742.2003. PMID 12574402
- [Result] Horger BA, Iyasere CA, Berhow MT, Messer CJ, Nestler EJ, Taylor JR. Enhancement of locomotor activity and conditioned reward to cocaine by brain-derived neurotrophic factor. J Neurosci. 1999 May 15;19(10):4110-22. doi: 10.1523/JNEUROSCI.19-10-04110.1999. PMID 10234039
- [Result] Jang EY, Yang CH, Hedges DM, Kim SP, Lee JY, Ekins TG, Garcia BT, Kim HY, Nelson AC, Kim NJ, Steffensen SC. The role of reactive oxygen species in methamphetamine self-administration and dopamine release in the nucleus accumbens. Addict Biol. 2017 Sep;22(5):1304-1315. doi: 10.1111/adb.12419. Epub 2016 Jul 14. PMID 27417190
- [Result] Ke X, Ding Y, Xu K, He H, Zhang M, Wang D, Deng X, Zhang X, Zhou C, Liu Y, Ning Y, Fan N. Serum brain-derived neurotrophic factor and nerve growth factor decreased in chronic ketamine abusers. Drug Alcohol Depend. 2014 Sep 1;142:290-4. doi: 10.1016/j.drugalcdep.2014.06.043. Epub 2014 Jul 11. PMID 25064020
- [Result] Khajebishak Y, Payahoo L, Alivand M, Alipour B. Punicic acid: A potential compound of pomegranate seed oil in Type 2 diabetes mellitus management. J Cell Physiol. 2019 Mar;234(3):2112-2120. doi: 10.1002/jcp.27556. Epub 2018 Oct 14. PMID 30317607
- [Result] Klintsova AY, Hamilton GF, Boschen KE. Long-term consequences of developmental alcohol exposure on brain structure and function: therapeutic benefits of physical activity. Brain Sci. 2012 Dec 21;3(1):1-38. doi: 10.3390/brainsci3010001. PMID 24961305
- [Result] Kovacic P. Role of oxidative metabolites of cocaine in toxicity and addiction: oxidative stress and electron transfer. Med Hypotheses. 2005;64(2):350-6. doi: 10.1016/j.mehy.2004.06.028. PMID 15607570
- [Result] Knaepen K, Goekint M, Heyman EM, Meeusen R. Neuroplasticity - exercise-induced response of peripheral brain-derived neurotrophic factor: a systematic review of experimental studies in human subjects. Sports Med. 2010 Sep 1;40(9):765-801. doi: 10.2165/11534530-000000000-00000. PMID 20726622
- [Result] Lange C, Storkebaum E, de Almodovar CR, Dewerchin M, Carmeliet P. Vascular endothelial growth factor: a neurovascular target in neurological diseases. Nat Rev Neurol. 2016 Aug;12(8):439-54. doi: 10.1038/nrneurol.2016.88. Epub 2016 Jul 1. PMID 27364743
- [Result] Misztak P, Panczyszyn-Trzewik P, Nowak G, Sowa-Kucma M. Epigenetic marks and their relationship with BDNF in the brain of suicide victims. PLoS One. 2020 Sep 24;15(9):e0239335. doi: 10.1371/journal.pone.0239335. eCollection 2020. PMID 32970734
- [Result] Mizrahi M, Friedman-Levi Y, Larush L, Frid K, Binyamin O, Dori D, Fainstein N, Ovadia H, Ben-Hur T, Magdassi S, Gabizon R. Pomegranate seed oil nanoemulsions for the prevention and treatment of neurodegenerative diseases: the case of genetic CJD. Nanomedicine. 2014 Aug;10(6):1353-63. doi: 10.1016/j.nano.2014.03.015. Epub 2014 Apr 2. PMID 24704590
- [Result] Novak G, LeBlanc M, Zai C, Shaikh S, Renou J, DeLuca V, Bulgin N, Kennedy JL, Le Foll B. Association of polymorphisms in the BDNF, DRD1 and DRD3 genes with tobacco smoking in schizophrenia. Ann Hum Genet. 2010 Jul;74(4):291-8. doi: 10.1111/j.1469-1809.2010.00578.x. Epub 2010 Apr 25. PMID 20456319
- [Result] Jeanblanc J, He DY, McGough NN, Logrip ML, Phamluong K, Janak PH, Ron D. The dopamine D3 receptor is part of a homeostatic pathway regulating ethanol consumption. J Neurosci. 2006 Feb 1;26(5):1457-64. doi: 10.1523/JNEUROSCI.3786-05.2006. PMID 16452669
- [Result] Ornell F, Hansen F, Schuch FB, Pezzini Rebelatto F, Tavares AL, Scherer JN, Valerio AG, Pechansky F, Paim Kessler FH, von Diemen L. Brain-derived neurotrophic factor in substance use disorders: A systematic review and meta-analysis. Drug Alcohol Depend. 2018 Dec 1;193:91-103. doi: 10.1016/j.drugalcdep.2018.08.036. Epub 2018 Oct 12. PMID 30347311
- [Result] Petrou P, Ginzberg A, Binyamin O, Karussis D. Beneficial effects of a nano formulation of pomegranate seed oil, GranaGard, on the cognitive function of multiple sclerosis patients. Mult Scler Relat Disord. 2021 Sep;54:103103. doi: 10.1016/j.msard.2021.103103. Epub 2021 Jun 27. PMID 34243101
- [Result] Qubty D, Frid K, Har-Even M, Rubovitch V, Gabizon R, Pick CG. Nano-PSO Administration Attenuates Cognitive and Neuronal Deficits Resulting from Traumatic Brain Injury. Molecules. 2022 Apr 23;27(9):2725. doi: 10.3390/molecules27092725. PMID 35566074
- [Result] Radak Z, Toldy A, Szabo Z, Siamilis S, Nyakas C, Silye G, Jakus J, Goto S. The effects of training and detraining on memory, neurotrophins and oxidative stress markers in rat brain. Neurochem Int. 2006 Sep;49(4):387-92. doi: 10.1016/j.neuint.2006.02.004. Epub 2006 Mar 27. PMID 16564605
- [Result] Requena-Ocana N, Flores-Lopez M, Papaseit E, Garcia-Marchena N, Ruiz JJ, Ortega-Pinazo J, Serrano A, Pavon-Moron FJ, Farre M, Suarez J, Rodriguez de Fonseca F, Araos P. Vascular Endothelial Growth Factor as a Potential Biomarker of Neuroinflammation and Frontal Cognitive Impairment in Patients with Alcohol Use Disorder. Biomedicines. 2022 Apr 20;10(5):947. doi: 10.3390/biomedicines10050947. PMID 35625687
- [Result] Skrabalova J, Drastichova Z, Novotny J. Morphine as a Potential Oxidative Stress-Causing Agent. Mini Rev Org Chem. 2013 Nov;10(4):367-372. doi: 10.2174/1570193X113106660031. PMID 24376392
- [Result] Tammela T, Enholm B, Alitalo K, Paavonen K. The biology of vascular endothelial growth factors. Cardiovasc Res. 2005 Feb 15;65(3):550-63. doi: 10.1016/j.cardiores.2004.12.002. PMID 15664381
- [Result] Turowski P, Kenny BA. The blood-brain barrier and methamphetamine: open sesame? Front Neurosci. 2015 May 5;9:156. doi: 10.3389/fnins.2015.00156. eCollection 2015. PMID 25999807
- [Result] Volkow ND, Koob G, Baler R. Biomarkers in substance use disorders. ACS Chem Neurosci. 2015 Apr 15;6(4):522-5. doi: 10.1021/acschemneuro.5b00067. Epub 2015 Mar 18. PMID 25734247
- [Result] Wan L, Xie Y, Su L, Liu Y, Wang Y, Wang Z. RACK1 affects morphine reward via BDNF. Brain Res. 2011 Oct 6;1416:26-34. doi: 10.1016/j.brainres.2011.07.045. Epub 2011 Jul 28. PMID 21885037
- [Result] Zamora-Lopez K, Noriega LG, Estanes-Hernandez A, Escalona-Nandez I, Tobon-Cornejo S, Tovar AR, Barbero-Becerra V, Perez-Monter C. Punica granatum L.-derived omega-5 nanoemulsion improves hepatic steatosis in mice fed a high fat diet by increasing fatty acid utilization in hepatocytes. Sci Rep. 2020 Sep 17;10(1):15229. doi: 10.1038/s41598-020-71878-y. PMID 32943651
- [Result] Zou Z, Wang H, d'Oleire Uquillas F, Wang X, Ding J, Chen H. Definition of Substance and Non-substance Addiction. Adv Exp Med Biol. 2017;1010:21-41. doi: 10.1007/978-981-10-5562-1_2. PMID 29098666